CLINICAL TRIAL: NCT01246570
Title: Supported Home-based Exercise Training Versus Usual Care After Cardiac Rehabilitation. A Randomized Controlled Study
Brief Title: Exercise Training Adherence After Cardiac Rehabilitation in Coronary Heart Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Adherence
Record Dates: First submitted 2010-11-16; First posted 2010-11-23 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Coronary Disease
Keywords: exercise; heart; coronary disease; rehabilitation
MeSH Terms: conditions — Coronary Disease; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Maintenance program (Experimental): Patients will attend a "motivational exercise session" once monthly. They will also be tested (exercise test with measurement of peak oxygen uptake) every third months.
  Interventions: Behavioral: Exercise training
- Control (Active Comparator): Usual care. The patients will receive the usual care provided by the hospital and community health services
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Exercise training — The patients will meet for organized exercise training once monthly and also exercise testing every third month.
  Arms: Maintenance program
Other: Control — The patients will receive the usual care provided by the hospitals and the community health services
  Arms: Control

SUMMARY:
It is known that organized cardiac rehabilitation is effective in improving exercise capacity in coronary heart disease patients. Less is known about the long-term results after cardiac rehabilitation. Earlier studies have shown that many patients quit exercising when no longer attending formal rehabilitation. The investigators wish to investigate the effect of a maintenance program after ending a rehabilitation program, and to compare this to usual care. The investigators hypothesis is that the maintenance program will result in higher exercise capacity and more physical activity compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* coronary heart disease patients

Exclusion Criteria:

* unstable angina pectoris
* hemodynamic significant valve disease (> New York Heart Association class II)
* pregnancy
* left ventricular ejection fraction <30%
* kidney failure (creatinin > 140)
* uncontrolled hypertension

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-11; Primary Completion 2013-04 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Peak oxygen uptake | baseline and 12 months
  The change in peak oxygen uptake from baseline to 12 months after baseline. In the intervention group, the peak oxygen uptake will be measured also every 3 months during the intervention period, and this will be reported

SECONDARY OUTCOMES:
Myocardial infarction | baseline and 12 months
  Diagnosis of myocardial infarction during the intervention period will be recorded
Hospital readmission | baseline and 12 months
  It will be recorded whether the patients is readmitted to hospital during the intervention period
Death | baseline and 12 months
Endothelial function | baseline and 12 months
  Flow mediated dilatation of the brachial artery, measured by ultrasound. Changes in flow-mediated dilatation from baseline to 12 months after baseline will be recorded
Quality of life | baseline and 12 months
  Mac New health related quality of life questionnaire. Changes in quality of life from baseline to 12 months after baseline will be recorded
Blood markers | baseline and 12 months
  Lipoproteins, c-peptide, ferritin, glucose, high sensitive c-reactive protein will be analysed. Also, blood will be stored for later analyses not yet planned. Changes in markers from baseline to 12 months after baseline will be recorded
Physical activity | baseline and 12 months
  Questionnaire and physical activity sensor (armband) will be measured at baseline and after 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Trine Moholdt, Phd, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway

REFERENCES:
- [Result] Madssen E, Arbo I, Granoien I, Walderhaug L, Moholdt T. Peak oxygen uptake after cardiac rehabilitation: a randomized controlled trial of a 12-month maintenance program versus usual care. PLoS One. 2014 Sep 23;9(9):e107924. doi: 10.1371/journal.pone.0107924. eCollection 2014. PMID 25247991